CLINICAL TRIAL: NCT05203692
Title: A Phase 1, Subjects- and Investigator-Blinded, Sponsor-Unblinded, Placebo-Controlled, Randomized, Sequential Cohort Study to Assess the Safety, Pharmacokinetics, and Pharmacodynamics of Single Ascending Intravenous and Subcutaneous Doses of DS-7011a in Healthy Subjects
Brief Title: A Study of a Single Ascending Dose Study of DS-7011a in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Daiichi Sankyo (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: DS7011-A-U101
Record Dates: First submitted 2022-01-20; First posted 2022-01-24 (Actual); Last update posted 2023-04-11 (Actual); Status verified 2023-04

CONDITIONS: Systemic Lupus Erythematosus
Keywords: Systemic Lupus Erythematosus; DS-7011a
MeSH Terms: conditions — Lupus Erythematosus, Systemic

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- DS-7011a (Experimental): Stage 1: Healthy participants who will be randomized to receive a single intravenous (IV) ascending dose of DS-7011a (starting dose 0.1 mg/kg).
  Stage 2: Healthy participants who will be randomized to receive a single subcutaneous (SC) ascending dose of DS-7011a (starting dose will be centered around estimated therapeutic dose confirmed in Stage 1).
  Stage 3: Healthy Japanese participants who will be randomized to receive an IV dose of DS-7011a (based on estimated therapeutic dose confirmed in Stage 1).
  Interventions: Drug: DS-7011a
- Placebo (Placebo Comparator): Healthy participants who will be randomized to receive a single dose of placebo.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: DS-7011a — Intravenous or subcutaneous administration, single dose
  Arms: DS-7011a
Drug: Placebo — Intravenous or subcutaneous administration, single dose
  Arms: Placebo

SUMMARY:
This will be the first-in-human study designed to evaluate the safety, pharmacokinetics (PK), and pharmacodynamics (PD) of single ascending doses of DS-7011a in healthy participants.

DETAILED DESCRIPTION:
This study will assess the safety, PK, and PD properties of single ascending intravenous (IV) and subcutaneous (SC) doses of DS-7011a in healthy participants.

This study will be conducted in 3 stages:

* Stage 1 - single ascending IV dose cohorts of DS-7011a (ie, up to 6 dose levels will be assessed starting at 0.1 mg/kg);
* Stage 2 - single ascending SC cohorts of DS-7011a (ie, up to 3 dose levels centered around the estimated therapeutic dose confirmed in Stage 1 will be assessed); and
* Stage 3 - a single IV cohort of DS-7011a in healthy participants of Japanese ethnicity (ie, 1 dose level at the estimated therapeutic dose as confirmed in Stage 1 will be assessed).

ELIGIBILITY:
Inclusion Criteria:

* Male and female participants 18 to 45 years of age (inclusive), with a body mass index (BMI) of 18 kg/m^2 to 30 kg/m^2 (inclusive) at Screening.
* Participants fully vaccinated against COVID-19 per current CDC guidelines or recovered from prior SARS-CoV-2 infection.
* All women must have a negative serum pregnancy test at Screening and a negative urine pregnancy test on Day -1.
* Women of childbearing potential must agree to use 2 different means of nonhormonal contraceptive methods.
* Women of non-childbearing potential must be either:

  * Surgically sterile (ie, bilateral tubal ligation or removal of both ovaries and/or uterus at least 6 months prior to dosing) or
  * Naturally postmenopausal for at least 24 consecutive months prior to dosing, spontaneous cessation of menses, with a follicle-stimulating hormone (FSH) level at Screening of ≥40 mIU/mL.
* Men must be surgically sterile (vasectomy 3 months before the dose of study drug) or agree to use approved contraception in addition to having their female partner (if of childbearing potential) use another acceptable form of contraception at any time during the study and for a period of 90 days after the dose of the study drug.
* Males may not donate sperm during the study for a period of 90 days
* Participants must be in overall good health, with no history of immunological and other chronic disorders, even if in remission and not requiring treatment.
* Confirmed Japanese ethnicity (Stage 3 only)

Exclusion Criteria:

* History or current chronic lung disease including asthma, COPD, or heavy smoking of >10 pack years
* Previous or current treatment with systemic corticosteroids or any immunosuppressive agents
* Participants who have received a transfusion or any blood products within the last year prior to dosing
* Participants who have made a blood donation or have had a loss of blood ≥500 mL within 56 days prior to the dose of study drug
* Participants who consume more than 28 units of alcohol per week (1 unit of alcohol equals 1/2 pint of beer, 4 ounces of wine, or 1 ounce of spirits) or those participants who have a significant history of alcoholism or drug/chemical abuse within the last 2 years
* Participants with positive results on tests for drugs of abuse, cotinine, or alcohol at Screening and/or Day -1

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2022-02-02 (Actual); Primary Completion 2023-01-25 (Actual); Study Completion 2023-03-22 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Treatment-emergent Adverse Events Following Administration with DS-7011a in Healthy Participants | Screening (Day -28 to Day -7) up to Day 57 post-dose
  Treatment-emergent adverse events (TEAEs) are defined as new adverse events (AEs) that occur after the dose of study drug or as AEs that were present prior to the dose of study drug but which worsened in severity after the start of study drug.

SECONDARY OUTCOMES:
Pharmacokinetic Parameter Area Under the Concentration Curve Following Administration of DS-7011a in Healthy Participants | Stage 1 and 3: Pre-dose, end of infusion (EOI), and 1, 3, 6, 12, 24, 48, and 96 hours post-EOI, Days 8, 11, 15, 22, 29, 36, and 57; Stage 2: Pre-dose, and 1, 3, 6, 12, 24, 36, 48, 72, 96, 120, 144, 168 hours post-dose, Days 9-12, 15, 22, 29, 36, and 57
  Area under the plasma concentration-time curve up to time t (AUCt), area under the plasma concentration-time curve up to infinity (AUCinf), and the percentage of AUCinf based on extrapolation (AUCextrap) will be calculated using noncompartmental methods.
Pharmacokinetic Parameter Maximum Concentration Following Administration of DS-7011a in Healthy Participants | Stage 1 and 3: Pre-dose, end of infusion (EOI), and 1, 3, 6, 12, 24, 48, and 96 hours post-EOI, Days 8, 11, 15, 22, 29, 36, and 57; Stage 2: Pre-dose, and 1, 3, 6, 12, 24, 36, 48, 72, 96, 120, 144, 168 hours post-dose, Days 9-12, 15, 22, 29, 36, and 57
  Maximum concentration (Cmax) will be calculated using noncompartmental methods.
Pharmacokinetic Parameter Time to Reach Maximum Plasma Concentration Following Administration of DS-7011a in Healthy Participants | Stage 1 and 3: Pre-dose, end of infusion (EOI), and 1, 3, 6, 12, 24, 48, and 96 hours post-EOI, Days 8, 11, 15, 22, 29, 36, and 57; Stage 2: Pre-dose, and 1, 3, 6, 12, 24, 36, 48, 72, 96, 120, 144, 168 hours post-dose, Days 9-12, 15, 22, 29, 36, and 57
  Time to reach maximum plasma concentration (Tmax) will be calculated using noncompartmental methods.
Pharmacokinetic Parameter Terminal Half-life Following Administration of DS-7011a in Healthy Participants | Stage 1 and 3: Pre-dose, end of infusion (EOI), and 1, 3, 6, 12, 24, 48, and 96 hours post-EOI, Days 8, 11, 15, 22, 29, 36, and 57; Stage 2: Pre-dose, and 1, 3, 6, 12, 24, 36, 48, 72, 96, 120, 144, 168 hours post-dose, Days 9-12, 15, 22, 29, 36, and 57
  Terminal half-life (t1/2) will be calculated using noncompartmental methods.
Mean Interleukin (IL)-6 Levels Following Administration of DS-7011a in Healthy Participants | Stage 1 and 3: Pre-dose, end of infusion (EOI), and 1, 3, 6, 12, 24, 48, and 96 hours post-EOI, Days 8, 11, 15, 22, 29, 36, and 57; Stage 2: Pre-dose, and 1, 3, 6, 12, 24, 36, 48, 72, 96, 120, 144, 168 hours post-dose, Days 9-12, 15, 22, 29, 36, and 57
  Mean IL-6 levels in whole blood stimulations will be assessed using ligand-activated toll-like receptor (TLR7) which stimulates IL-6 production.
Proportion of Participants Who Are Anti-Drug Antibody (ADA)-Positive (Baseline and Post-Baseline) and Proportion of Participants Who Have Treatment-emergent ADA | Pre-dose (Day 1) up to Day 57 post-dose

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Leader, Study Director — Daiichi Sankyo
Locations (2):
- United States (2):
  - Apex Clinical Research (Collaborative Neuroscience Research), Long Beach, California
  - Worldwide Clinical Trials, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: No